CLINICAL TRIAL: NCT06772545
Title: A Prospective Comparative Study on the Effects of Multimodal Analgesia Regimens on Postoperative Analgesia and Gastrointestinal Function Recovery After Laparoscopic Abdominal Surgery
Brief Title: Study on the Effects of Multimodal Analgesia Regimens on Postoperative Analgesia and Gastrointestinal Function Recovery After Laparoscopic Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-321
Record Dates: First submitted 2025-01-10; First posted 2025-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Laparoscopic Abdominal Surgery
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- EA (Experimental): Epidural Analgesia
  Interventions: Procedure: Epidural Analgesia
- PB (Experimental): Paravertebral Block
  Interventions: Device: Paravertebral Block
- TAP (Experimental): Transversus Abdominis Plane Block
  Interventions: Device: Transversus Abdominis Plane Block
- PCIA (Active Comparator): Patient-Controlled Intravenous Analgesia
  Interventions: Device: patient-controlled intravenous analgesia (PCA)

INTERVENTIONS:
Procedure: Epidural Analgesia — Patients in the EA group underwent epidural anesthesia after admission to the operating room. Following successful epidural puncture, 3 ml of 2% lidocaine was administered. Once the block level was confirmed, the epidural analgesia pump was activated, delivering 8 ml/h of 0.1% ropivacaine.
  Arms: EA
Device: Paravertebral Block — Using an in-plane technique, the puncture needle was advanced from lateral to medial under real-time ultrasound guidance to the target paravertebral space, passing through the intercostal fascia, avoiding the parietal pleura, and positioning the needle tip superior to the costotransverse ligament. After confirming needle tip placement, 10 mL of 0.5% ropivacaine was slowly injected in divided doses, observing for the spread of the local anesthetic to ensure adequate distribution within the PVS for effective block.
  Arms: PB
Device: Transversus Abdominis Plane Block — The plane of blockade and whether to perform a single or double injection technique were determined based on the incision location. Under real-time ultrasound guidance, the puncture needle was advanced to the target transversus abdominis plane. After confirming needle tip placement, 10 mL of 0.5% ropivacaine was injected slowly in a fractionated manner while observing the local anesthetic spread to ensure effective blockade.
  Arms: TAP
Device: patient-controlled intravenous analgesia (PCA) — The patient-controlled analgesia (PCA) device was programmed to deliver bolus doses of 15 μg fentanyl, with a 10-minute lockout period and no background infusion. The PCA solution consisted of 1 mg fentanyl and 8 mg of tropisetron mixed in 100 mL of normal saline.
  Arms: PCIA

SUMMARY:
This clinical trial aims to investigate the impact of multimodal analgesia regimens on postoperative pain management and gastrointestinal function recovery following laparoscopic abdominal surgery. The primary objectives are to determine:

Which analgesic regimen is most effective in reducing postoperative pain? Which analgesic regimen is most effective in accelerating gastrointestinal function recovery? This study will compare epidural analgesia (EA), paravertebral block (PB), transversus abdominis plane block (TAP), and patient-controlled intravenous analgesia (PCIA) to identify the optimal method for pain control and the most beneficial for gastrointestinal recovery.

Participants will receive one of the following treatments postoperatively: epidural analgesia, paravertebral block, TAP block, or patient-controlled intravenous analgesia. Rest pain (measured using the Numerical Rating Scale, NRS), dynamic pain (NRS), morphine equivalent consumption (mg), quality of sleep on the first night (Likert scale, 1-5), time to return of bowel function (h), time to recommence oral intake (h), time to first mobilization (h), quality of recovery (QoR, 0-15) on postoperative day 1, and length of hospital stay (days) will be recorded at 4, 8, 12, and 24 hours post-procedure.

DETAILED DESCRIPTION:
Study design：This is a prospective, randomized, comparative, double-blind study designed to assess the superiority and non-inferiority of four analgesic techniques: epidural analgesia (EA), paravertebral block (PB), transversus abdominis plane block (TAP), and patient-controlled intravenous analgesia (PCIA). The study will evaluate the effectiveness of these methods for pain management in patients undergoing laparoscopic abdominal surgery. Patients will be recruited at Baogang Hospital in Inner Mongolia. This study was approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia, and adhered to the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed consent voluntarily.

Patients：A total of 120 patients undergoing laparoscopic abdominal surgery, classified as American Society of Anesthesiologists (ASA) physical status I-III, will be recruited between February and May 2025. These patients will be randomly assigned to one of four groups, with 30 patients in each group. Randomization and Blinding：This study employed block randomization to generate the random allocation sequence. A block size of 6 was set, and the random sequence was generated using dedicated software (the blockrand package in R version 4.3.2). The allocation of the random sequence was performed by an independent third party, and allocation concealment was implemented using sequentially numbered, sealed, opaque envelopes. The research team remained blinded throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention： General anesthesia and monitoring Upon arrival in the operating room, patients were monitored for pulse oximetry (SPO2), electrocardiogram (ECG), bispectral index (BIS), and non-invasive arterial blood pressure. Pain threshold (PTh, mA) and pain tolerance threshold (PTTh, mA) were measured and recorded. Patients received pre-operative administration of Penehyclidine Hydrochloride Injection (Lot H20051948, Chengdu List Pharmaceutical Co., Ltd., China) (0.01 mg kg-1 i.v.). Induction was achieved with propofol (1.5-2 mg kg-1 i.v.), rocuronium bromide (1-2 mg kg-1 i.v.), and fentanyl (1-2 μg kg-1 i.v.). Anesthesia was maintained with inhaled sevoflurane or desflurane, with the inhaled concentration adjusted according to BIS values. Remifentanil (0.05-0.2 μg kg-1 min-1 i.v.) was continuously infused to maintain blood pressure and heart rate within ±20% of baseline values. Mechanical ventilation was initiated in pressure-regulated volume control (PRVC) mode after induction. Ventilator settings (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) were as follows: tidal volume 6-8 ml kg-1, positive end-expiratory pressure (PEEP) 0 cmH2O, inspiratory-to-expiratory ratio 1:2, respiratory rate 16 beats per minute (BPM), and inspired oxygen concentration 41%. The patient was positioned in the Trendelenburg position, with the operating table tilted 20-25° head down. Carbon dioxide pneumoperitoneum was established at an intra-abdominal pressure of 10-15 mmHg.

Postoperative care Vital signs were monitored in the Post Anesthesia Care Unit (PACU), with supplemental oxygen provided via facemask. For hypotension, ephedrine (6-10 mg) was administered, and fluid administration was increased. Atropine (0.3-0.5 mg) was given for bradycardia. For pain, sufentanil (0.1-0.2 μg/kg) was administered.

Data collection Upon arrival in the operating room, heart rate (HR, bpm), mean arterial pressure (MAP, mmHg) (calculated as MAP = diastolic pressure + 1/3 pulse pressure), BIS, remifentanil dosage (mg), ephedrine dosage (mg), duration of surgery (minutes), and duration of anesthesia (minutes) were recorded for all patients.

In the PACU, the following data were recorded: number of patients requiring sufentanil (μg), number of patients experiencing respiratory depression (n), number of hypotension events requiring intervention (n), ephedrine dosage (mg), intravenous fluid volume (ml), number of patients experiencing bradycardia (n), atropine dosage (mg), Bromage score, and time spent in the PACU (min). For patients transferred to the high dependency unit, the number of patients (n) and length of stay (h) were recorded.

Postoperatively, rest pain (Numerical Rating Scale, NRS), dynamic pain (NRS), morphine equivalent (mg), quality of sleep on the first night (Likert scale, 1-5), functional recovery (return of bowel function, h, recommencement of oral intake, h, and time to first mobilization, h), quality of recovery (QoR, 0-15) on postoperative day 1, and hospital stay (days) were recorded at 4, 8, 12, and 24 hours. Ketorolac dosage (mg), hydromorphone dosage (mg), oral medications, number of episodes of PONV (n), antiemetic dosage (mg), number of episodes of pruritus (n), and Comprehensive Complication Index (CCI) were recorded over 24 hours.

Outcomes and measures：Patient follow-up was conducted in the ward by two specially trained nurses who were blinded to patient group assignment. Assessments, including those for postoperative day 1 and length of hospital stay, were performed in person at 4, 8, 12, and 24 hours post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* ASA I-III
* Ability to understand and voluntarily sign the informed consent form
* No prior use of long-acting or addictive analgesic drugs before surgery.

Exclusion Criteria:

* History of previous abdominal surgery
* Presence of severe cardiovascular, respiratory, hepatic, renal, neurological, or psychiatric disorders
* Pre-existing chronic pain conditions
* Known allergy to any analgesic drugs used in this study
* Presence of spinal deformities, neurological conditions, or coagulopathy that may affect the performance of regional anesthesia.
* Pregnant or breastfeeding women
* Inability to cooperate with study procedures or understand pain rating scales
* History of opioid abuse or addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | at 4 hours post-treatment, 8 hours post-treatment, 12 hours post-treatment, and 24 hours post-treatment
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Functional recovery Return bowel function(h) | At 72 hours post-surgery
  A participant was considered to have achieved a response if their performance status score was either 0 or 72 hours, on a scale where 0 represented the best outcome and 72 the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Wang, MM, Principal Investigator — Inner Mongolia Baogang Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2036
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.